CLINICAL TRIAL: NCT04568941
Title: Randomized Controlled Trial of Comparison of Tumor Biopsy Method of Preoperative Vacuum-Assisted, Core Needle Versus Intraoperative Excisional Biopsy for Sentinel Lymph Node Biopsy in Breast Cancer
Brief Title: Comparison Study of Different Tumor Biopsy Method for Sentinel Lymph Node Biopsy in Breast Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shandong Cancer Hospital and Institute (Other)
Responsible Party: Principal Investigator, Zhiyong Yu, Zhiyong Yu, Shandong Cancer Hospital and Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ShandongCHI-13
Record Dates: First submitted 2020-09-26; First posted 2020-09-29 (Actual); Last update posted 2020-10-27 (Actual); Status verified 2020-10

CONDITIONS: Breast Cancer; Sentinel Lymph Node
Keywords: Sentinel Lymph Node; vacuum-assisted biopsy; Core needle biopsy; Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Biopsy, Large-Core Needle

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Preoperative Vacuum-Assisted Biopsy (Experimental): Preoperative vacuum-assisted biopsy was performed within 10 days before final surgery. The tumor were excised almost.
  Interventions: Behavioral: Vacuum-Assisted Biopsy
- Preoperative Core Needle Biopsy (Experimental): Preoperative core needle biopsy was performed within 10 days before final surgery. The needle biopsy were performed with 3 needles.
  Interventions: Behavioral: Core Needle Biopsy
- Intraoperative Excisional Biopsy (Experimental): The tumor was excised intraoperatively.
  Interventions: Behavioral: Intraoperative Excisional Biopsy

INTERVENTIONS:
Behavioral: Vacuum-Assisted Biopsy — Vacuum-Assisted Biopsy
  Arms: Preoperative Vacuum-Assisted Biopsy
Behavioral: Core Needle Biopsy — Core Needle Biopsy
  Arms: Preoperative Core Needle Biopsy
Behavioral: Intraoperative Excisional Biopsy — Intraoperative Excisional Biopsy
  Arms: Intraoperative Excisional Biopsy

SUMMARY:
Sentinel lymph node biopsy (SLNB) has become a mainstay surgery method in breast cance, and the identified number of sentinel lymph nodes determines its accuracy for axillary status. Retrospective study indicated that preoperative tumor biopsy results in more detected sentinel lymoh nodes. The clinical trail is designed to compare the effect of three tumor biopsy methods (preoperative vacuum-assisted biopsy, core needle biopsy, and intraoperative excisional biopsy) for sentinel lymph nodes.

DETAILED DESCRIPTION:
OBJECTIVES:

Compare the identification rate of sentinel lymph node in breast cancer patients with different tumor biopsy methods.

Evaluate the false-negative rates of sentinel lymph nodes in patients with different tumor biopsy methods.

OUTLINE:

The patients were randomly divided into three group, vacuum-assisted biopsy, core needle biopsy, and intraoperative excisional biopsy. Preoperative vacuum-assisted biopsy and core needle biopsy were performed in 10 days before the final surgery. All patients received dual tracer (radiolabeled colloid and blue dye) guided SLNB.

ELIGIBILITY:
Inclusion Criteria:

* clinically lymph node negative breast cancer patients T1-T3

Exclusion Criteria:

* history of breast cancer locally advanced breast cancer and metastatic breast cancer proven axillary lymph node metastasis history of axillary excisional or incisional biopsy, or dissection history of neoadjuvant chemotherapy pregnancy non-consented patients

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2020-11-01 (Estimated); Primary Completion 2021-05-01 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
Identification rates of sentinel lymph node biopsy | 1 year
  Identification rate of SLNB between three groups

SECONDARY OUTCOMES:
Identification numbers of sentinel lymph node biopsy | 1 year
  Identification numbers of SLNB between three groups
fase-negative rates of sentinel lymph node biopsy | 1 year
  fase-negative rates of SLNB between three groups

CONTACTS AND LOCATIONS:
Locations (1):
- Zhiyong Yu, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Yuan C, Wang X, Liu Z, Li C, Bian M, Shan J, Song X, Yu Z, Yu J. Preoperative tumor biopsy results in more detected sentinel nodes than intraoperative biopsy in breast cancer patients. World J Surg Oncol. 2020 Jul 21;18(1):178. doi: 10.1186/s12957-020-01942-4. PMID 32693797
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/32693797/